CLINICAL TRIAL: NCT06882655
Title: A Combination of Intrathecal Fentanyl and Ultrasound-Guided Pecto-Intercostal Fascial Block in Paediatric Cardiac Surgery: A Randomized Controlled Trial
Brief Title: A Combination of Intrathecal Fentanyl and Pecto-Intercostal Fascial Block in Paediatric Cardiac Surgery.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB NO : 00012098
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Pain; Pediatric Open Heart Surgery
Keywords: Intercostal Fascial Block; intrathecal fentanyl; Paediatric Cardiac Surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pecto-Intercostal Fascial Block group (Experimental): The PIFB group (Group PIFB; n = 30) will receive a pecto-intercostal-fascial plane block (PIFB). The blocks will be performed bilaterally in a supine position after induction of anaesthesia. The in-plane needle approach will be applied under the guidance of a high-frequency Hockey Stick Linear-Array US transducer probe (SONOSITE M-TURBO). Under strict aseptic precautions, the transducer will be placed 1-2 cm lateral to and parallel to the sternum to count the ribs from the second to the sixth rib. A 22-gauge, 50-mm short bevel echogenic needle will be advanced in a caudal-to-cranial direction until the tip of the needle will be in the targeted fascial plane, a test bolus of normal saline (1-2 mL) will be injected (in real-time) to confirm that the tip was correctly placed, as shown by separation of the fascial layers. After excluding intravascular, the dose of local anaesthetic (0.4 mL/kg 0.25% bupivacaine) will be deposited into the fascial plane visualised in real-time.
  Interventions: Procedure: PIFB group
- Intrathecal fentanyl group (Active Comparator): The children in the IT fentanyl group (Group IT; n = 30) will be placed in lateral decubitus position immediately after intubation and catheterisation and receive an IT injection of 2 µg/kg of fentanyl in 0.2 mL/kg of normal saline through a 2-in., 25-gauge Quincke spinal needle inserted at L3-4 or L4-5. The dose of IT fentanyl will be based on a previous study. (15) with this route of fentanyl administration to provide intraoperative analgesia and blunt the stress response in pediatric cardiac anaesthesia. Successful dural puncture will be confirmed by observation of a free flow of cerebrospinal fluid, and the injection will be performed with the bevel of the needle oriented in the cephalic direction.
  Interventions: Procedure: Intrathecal fentanyl(IT fentanyl)
- intrathecal fentanyl and pectointercostal fascial block (Active Comparator): Patients assigned to the combined IT fentanyl and PIFB (Group IT + PIFB; n = 30) will receive both a PIFB and IT fentanyl, with the use of the methods described for the other two groups.
  Interventions: Procedure: IT + PIFB

INTERVENTIONS:
Procedure: PIFB group — A pecto-intercostal-fascial plane block (PIFB) will be performed bilaterally in a supine position after induction of anaesthesia. The in-plane needle approach will be applied under the guidance of a high-frequency Hockey Stick Linear-Array US transducer probe (SONOSITE M-TURBO). Under strict aseptic precautions, the transducer will be placed 1-2 cm lateral to and parallel to the sternum to count the ribs from the second to the sixth rib. A 22-gauge, 50-mm short bevel echogenic needle will be advanced in a caudal-to-cranial direction until the tip of the needle will be in the targeted fascial plane, a test bolus of normal saline (1-2 mL) will be injected (in real-time) to confirm that the tip was correctly placed, as shown by separation of the fascial layers. After excluding intravascular, the dose of local anaesthetic (0.4 mL/kg 0.25% bupivacaine) will be deposited into the fascial plane visualised in real-time.
  Arms: Pecto-Intercostal Fascial Block group
Procedure: Intrathecal fentanyl(IT fentanyl) — IT fentanyl group (Group IT; n = 30) will be placed in lateral decubitus position immediately after intubation and catheterisation and receive an IT injection of 2 µg/kg of fentanyl in 0.2 mL/kg of normal saline through a 2-in., 25-gauge Quincke spinal needle inserted at L3-4 or L4-5. The dose of IT fentanyl will be based on a previous study. (15) with this route of fentanyl administration to provide intraoperative analgesia and blunt the stress response in pediatric cardiac anaesthesia. Successful dural puncture will be confirmed by observation of a free flow of cerebrospinal fluid, and the injection will be performed with the bevel of the needle oriented in the cephalic direction.
  Arms: Intrathecal fentanyl group
Procedure: IT + PIFB — Patients assigned to the combined IT fentanyl and PIFB (Group IT + PIFB; n = 30) will receive both a PIFB and IT fentanyl, with the use of the methods described for the other two groups.
  Arms: intrathecal fentanyl and pectointercostal fascial block

SUMMARY:
Cardiac surgery is commonly performed via median sternotomy. Patients undergoing cardiac surgical procedures frequently experience intense acute pain in the post-sternotomy wound, which can potentially transition into persistent chronic pain in approximately 35% of cases after one year. Recently, thoracic myofascial plane blocks with ultrasound guidance as part of multimodal analgesia have contributed to a faster recovery after surgery.

De la Torre et al. first described pectointercostal fascial plane block (PIFPB) for breast surgery. Local anaesthetics are injected between the pectoralis major and internal intercostal muscles close to the sternum to block the anterior cutaneous branch of the second-to-sixth thoracic intercostal nerves.The use of intrathecal (IT) opioids with or without local anaesthetics (LA) is a popular analgesic technique around the world for the management of postoperative pain. Unlike IT administration of LA, IT opioids produce 'segmental' analgesia and are not associated with muscle weakness, loss of proprioception or sympathetic block. IT opioids can be administered as an adjunct to general anaesthesia or combined with LA and administered during spinal anaesthesia for surgery. It is one of the easiest, most reliable and cost-effective methods for pain relief. Intrathecal opioid administration can provide more intense analgesia than the IV route and has the advantages of simplicity and reliability

DETAILED DESCRIPTION:
Cardiac surgery is commonly performed via median sternotomy. Patients undergoing cardiac surgical procedures frequently experience intense acute pain in the post-sternotomy wound, which can potentially transition into persistent chronic pain in approximately 35% of cases after one year. Sternal wound pain has been linked to diminished patient satisfaction, delirium, and a spectrum of cardiovascular complications, including hypotension, tachycardia, arrhythmias, and respiratory issues such as stasis of bronchial secretions, atelectasis, and pneumonia.

Pain management after cardiac surgery is critical to enhancing recovery. Various modalities are available for managing postoperative pain in cardiac surgery. These modalities include opioids, local anaesthetic techniques such as local anaesthetic infiltration, and neuraxial blocks (epidural and paravertebral). Additionally, acetaminophen and nonsteroidal anti-inflammatory drugs (NSAIDs) are feasible options for pain control. Furthermore, adjunct analgesics such as steroids, ketamine, α2 agonists, and anticonvulsants are also employed for effective pain management.Opioids can elicit various adverse effects, such as delayed tracheal extubation, respiratory depression, sedation, ileus, nausea, vomiting, immunosuppression, cough suppression, drowsiness, and an increased risk of chronic pain.

Recently, thoracic myofascial plane blocks with ultrasound guidance as part of multimodal analgesia have contributed to a faster recovery after surgery.

De la Torre et al.first described pectointercostal fascial plane block (PIFPB) for breast surgery. Local anaesthetics are injected between the pectoralis major and internal intercostal muscles close to the sternum to block the anterior cutaneous branch of the second-to-sixth thoracic intercostal nerves. PIFPB has been an effective technique for pain control after sternotomy . However, a high incidence of non-sternal wound pain was observed with this technique of fascial plain block both in adults and paediatrics after cardiac surgery .

The use of intrathecal (IT) opioids with or without local anaesthetics (LA) is a popular analgesic technique around the world for the management of postoperative pain. Unlike IT administration of LA, IT opioids produce 'segmental' analgesia and are not associated with muscle weakness, loss of proprioception or sympathetic block. IT opioids can be administered as an adjunct to general anaesthesia or combined with LA and administered during spinal anaesthesia for surgery. It is one of the easiest, most reliable and cost-effective methods for pain relief. Intrathecal opioid administration can provide more intense analgesia than the IV route and has the advantages of simplicity and reliability.

ELIGIBILITY:
Inclusion Criteria:

* The enrolled patients ranged in age from 6 months to 6 years,
* patients scheduled for surgical repair of congenital heart defects.

Exclusion Criteria:

* The preoperative criteria include a history of previous cardiac surgery, hemodynamic instability, the need for mechanical ventilation, and the requirement for vasoactive drugs, opioids, or corticosteroids.
* During the intraoperative phase, who use of deep hypothermic circulatory arrest and the necessity for vasoactive drugs, excluding the temporary use of dopamine and dobutamine at a maximum dose of 10 µg/kg/min.
* Postoperative exclusion conditions will include prolonged mechanical ventilation lasting more than 24 hours, hemodynamic instability, and the need for high doses of opioids or sedatives.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
To investigate how effectively three distinct pain management techniques can reduce the stress response that patients experience after undergoing cardiac surgery. | after the procedure24 hour
  Serum cortisol and plasma epinephrine and norepinephrine will be measured.

SECONDARY OUTCOMES:
To conduct a comparative analysis of the analgesic efficacy of each pain management method. | every 30 minutes for the first six postoperative hours and every 6 hours during the first, second, and third postoperative days.
  -Analgesia/sedation scores will be recorded The team will evaluate each child for the level of analgesia and sedation using the COMFORT scale. (16) (before extubation) and the Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) (17) (after extubation)
To meticulously document and evaluate any potential adverse effects associated with these pain management strategies, ensuring patient safety. | first 30 min after block administration and 24 hour postoperatively
  The incidence of adverse events associated with the block is as follows: local anaesthesia toxicity (neurologic or cardiovascular events occurring within the first 30 min after block administration), chest wall hematoma, and pneumothorax (diagnosed by the US after block and before skin incision).
to determine which technique offers the most effective in early extubation | in first 24 hour postoperatively
  The time to extubate (in minutes )
to determine the duration of analgesic effect of technique post operative | in first 24 hour postoperatively
  The time for first rescue analgesia in minutes
to determine which technique offers lesser consumption of fentanyl | intraoperative during the procedure and first 3 days post operative
  The total dose of fentanyl consumed intraoperatively and for each of the first 3 days postoperatively (µg/kg).

CONTACTS AND LOCATIONS:
Overall Officials: Islam Elbardan, Dr, Principal Investigator — University of Alexandria
Locations (1):
- Faculty of medicine ,Alexandria university, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No